CLINICAL TRIAL: NCT03221374
Title: Mind-body Awareness Training and Brain-computer Interface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Dr. Bin He, Professor of Biomedical Engineering, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R01AT009263-01 (NIH)
Record Dates: First submitted 2017-07-07; First posted 2017-07-18 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): Participants will attend an 8-week Mindfulness Based Stress Reduction (MBSR) course between pre- and post-testing.
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Waitlist (No Intervention): Participants will be added to a waitlist intervention group for 8-weeks between pre-and post-testing.

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — 8-week mindfulness based stress reduction course intended to develop mind-body awareness through mindfulness practices.
  Arms: Mindfulness Based Stress Reduction

SUMMARY:
Mind-Body Awareness Training (MBAT), in the forms of various yoga and meditative practices, has become increasingly prevalent due to an increase in awareness of the potential health benefits, and improvements in concentration that this training can provide to practitioners. In the present study, the role of Mind-Body Awareness Training (MBAT) in the initial learning of a sensorimotor (SMR) based Brain-Computer Interface (BCI) is being investigated. The hypothesis is that MBAT will improve performance in SMR based BCI.

DETAILED DESCRIPTION:
In this protocol, the following hypothesis will be tested; namely that MBAT including the verified mindfulness based stress reduction (MBSR) course will improve the ability for subjects to concentrate on the control of the SMR thus improving the performance of BCI. Subjects will be recruited for short term MBAT and then undergo BCI training. The performance of subjects with MBAT will be compared with those without MBAT to test the hypothesis. Procedures involved include a standard 8-week MBSR course, and an EEG brain noninvasive brain computer interface study.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy volunteers
* Age 18-64, inclusive.
* Willing and able to provide written consent.
* Able to communicate in the English language.

Exclusion Criteria:

* Any past BCI experience.
* Pregnancy
* Any breathing, movement, or visual disorders.
* Any active neurological or mental disorders.
* History of epilepsy.
* History of a vascular or cardiac disorder (e.g. heart disease)
* History of a metabolic disorder (e.g. diabetes)
* Any other condition which would make the subject, in the opinion of the investigator, unsuitable for the study.

Exclusion criteria that would prevent subjects from participating in the optional MRI component will be:

* Any MRI incompatible indwelling metal objects or implantable devices, including but not limited to the following (dental mental is allowable):

  * Cardiac pacemaker
  * Implanted cardiac defibrillator
  * Carotid artery vascular clamp
  * Intravascular stents, filters, or coils
  * Aortic clip
  * Internal pacing wires
  * Vascular access port and/or catheter
  * Swan-Ganz catheter
  * Shunt (spinal or intraventricular)
  * Aneurysm clip(s)
  * Neurostimulator
  * Electrodes (on body, head, or brain)
  * Heart valve prosthesis
  * Any type of prosthesis (eye, penile, etc.)
  * Artificial limb or joint replacement
  * Bone growth/fusion stimulator
  * Bone/joint pin, screw, nail, wire, plate
  * Metal rods in bones
  * Harrington rods (spine)
  * Metal or wire mesh implants
  * Wire sutures or surgical staples
  * Insulin pump or infusion device
  * Any metal fragments (i.e. metal shop)
  * Any implant held in place by a magnet
  * Cochlear, otologic, or ear implant
* Claustrophobia
* Hearing aid use
* Any yoga/meditation in the last three months.
* More than 12 yoga/meditation classes in the last 12 months.
* Approximately weekly yoga/meditation for a year or more at any point in the past.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 231 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bin He, Ph.D, Principal Investigator — Carnegie Mellon University
Locations (1):
- Biomedical Engineering Department Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by flyers posted around the campus, references by the meditator instructors, or department emails.
Pre-assignment Details: Subjects will be excluded, if they tell the experimenter that they do not wish to continue the participation.
Groups:
- Mindfulness Based Stress Reduction - UMN: Participants will attend an 8-week Mindfulness Based Stress Reduction (MBSR) course between pre- and post-testing. This cohort of experiment was performed at the University of Minnesota (UMN).
  Mindfulness Based Stress Reduction: 8-week mindfulness based stress reduction course intended to develop mind-body awareness through mindfulness practices.
- Waitlist - UMN: Participants will be added to a waitlist intervention group for 8-weeks between pre-and post-testing. This cohort of experiment was performed at the University of Minnesota (UMN).
- Experienced Meditator - CMU: Participants that have more than 1 year of regular meditation experience, and will perform a series of brain-computer interface experiments.
- Meditation Naive - CMU: Participants that have no regular meditation experience, and will perform a series of brain-computer interface experiments.
- Mindfulness Based Stress Reduction - CMU: Participants will attend an 8-week Mindfulness Based Stress Reduction (MBSR) course between pre- and post-testing. This cohort of experiment was performed at the Carnegie Mellon University (CMU).
  Mindfulness Based Stress Reduction: 8-week mindfulness based stress reduction course intended to develop mind-body awareness through mindfulness practices.
- Waitlist - CMU: Participants will be added to a waitlist intervention group for 8-weeks between pre-and post-testing. This cohort of experiment was performed at the Carnegie Mellon University (CMU).
- Short Term Meditation - CMU - Meditation: Participants will undergo a 20-minute meditation between two Brain-computer interface sessions.
- Short Term Meditation - CMU - Control: Participants will listen to a 20-min reading of meditation related journal article between two Brain-computer interface sessions.
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction - UMN | Waitlist - UMN | Experienced Meditator - CMU | Meditation Naive - CMU | Mindfulness Based Stress Reduction - CMU | Waitlist - CMU | Short Term Meditation - CMU - Meditation | Short Term Meditation - CMU - Control
Started | 72 | 72 | 32 | 34 | 8 | 8 | 3 | 2
Completed | 42 | 34 | 22 | 26 | 7 | 5 | 2 | 1
Not Completed | 30 | 38 | 10 | 8 | 1 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The population described here are participants enrolled in each arm/group, which is consistent with the participants flow section.
Groups:
- Mindfulness Based Stress Reduction - UMN; Mindfulness Based Stress Reduction - CMU: Participants will attend an 8-week Mindfulness Based Stress Reduction (MBSR) course between pre- and post-testing.
  Mindfulness Based Stress Reduction: 8-week mindfulness based stress reduction course intended to develop mind-body awareness through mindfulness practices.
- Waitlist - UMN; Waitlist - CMU: Participants will be added to a waitlist intervention group for 8-weeks between pre-and post-testing.
- Experienced Meditator - CMU: participants that have more than 1 year of regular meditation experience
- Meditation Naive - CMU: Participants that have no regular meditation experience
- Short Term Meditation - CMU - Control: Participants will listen to a 20-min reading of meditation related journal aritcle between two Brain-computer interface sessions.
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction - UMN | Waitlist - UMN | Experienced Meditator - CMU | Meditation Naive - CMU | Mindfulness Based Stress Reduction - CMU | Waitlist - CMU | Short Term Meditation - CMU - Meditation | Short Term Meditation - CMU - Control | Total
Number analyzed (Participants) | 72 | 72 | 32 | 34 | 8 | 8 | 3 | 2 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (14.6) | 34.1 (13.3) | 41.6 (16.5) | 26.5 (9.3) | 32.3 (15.4) | 26.8 (8.0) | 45.7 (19.3) | 39.5 (4.9) | 35.2 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 59 | 17 | 23 | 5 | 2 | 2 | 0 | 164
  Male | 16 | 13 | 15 | 11 | 3 | 6 | 1 | 2 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 6
  Not Hispanic or Latino | 63 | 63 | 30 | 30 | 7 | 8 | 3 | 2 | 206
  Unknown or Not Reported | 7 | 8 | 2 | 2 | 0 | 0 | 0 | 0 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 7 | 2 | 5 | 0 | 6 | 0 | 0 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 4 | 1 | 2 | 0 | 1 | 12
  White | 57 | 56 | 24 | 21 | 6 | 0 | 3 | 1 | 168
  More than one race | 7 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 10
  Unknown or Not Reported | 4 | 6 | 2 | 4 | 1 | 0 | 0 | 0 | 17
Prior regular meditation experience over 1 year [Count of Participants; unit: Participants] — This measure is about whether a participant has a regular meditation experience of over 1 year, which defines a participant as an experienced meditator.
  Participants | 0 | 0 | 32 | 0 | 0 | 0 | 1 | 0 | 33

OUTCOME MEASURES:

1. Primary Outcome: BCI Performance Change From Baseline
Description: This outcome is related to the sub-study to investigate the effect of the MBSR on BCI learning. During the course of the sub-study over approximately 6 months/cohort of participants, participant learning over time during the course of study will be examined in terms of performance change after the intervention as well as across sessions, with a positive number representing an increase, and a negative number to represent a decrease. The percent valid correct (percent correct over valid trials) metric will be used to evaluate learning.
Time Frame: 6 months for each participant.
Population: The population consists of participants recruited in the UMN site to investigate the effect of 8-week MBSR class on the effect of BCI learning. During the analysis, participants were excluded if they dropped the experiment, did not follow the task guideline, or exhibited ceiling performance.
  The number of participants in the "Mindfulness-Based Stress Reduction - CMU", "Waitlist - CMU" are too small to draw statistical conclusions and thus were not included.
Measure: Mean (Standard Deviation); unit: Percent valid correct (PVC)
Groups:
- Mindfulness Based Stress Reduction - UMN: Participants will attend an 8-week Mindfulness Based Stress Reduction (MBSR) course between pre- and post-testing. This cohort of experiment was performed at the Carnegie Mellon University (CMU).
  Mindfulness Based Stress Reduction: 8-week mindfulness based stress reduction course intended to develop mind-body awareness through mindfulness practices.
- Waitlist - UMN: Participants will be added to a waitlist intervention group for 8-weeks between pre-and post-testing. This cohort of experiment was performed at the Carnegie Mellon University (CMU).
Arm/Group | Mindfulness Based Stress Reduction - UMN | Waitlist - UMN
Number analyzed (Participants) | 33 | 29
Percent valid correct (PVC) | 16.87 (14.55) | 7.9 (15.96)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction - UMN vs Waitlist - UMN; Test type: Other — Linear mixed effect model to test the overall BCI learning between MBSR and control groups; p = 0.003, Mixed Models Analysis — The threshold for statistical analysis was p = 0.05
Statistical Analysis 2: Comparison: Mindfulness Based Stress Reduction - UMN vs Waitlist - UMN; Test type: Equivalence — This independent t-test will test if the two groups (MBSR, control) exhibit a statistically significant difference in terms of BCI performance from baseline; p = 0.024, t-test, 2 sided — The threshold for statistical analysis was p = 0.05; Mean Difference (Net) = 8.98 — The difference between BCI performance improvement in MBSR cohort and control cohort

2. Primary Outcome: Breath Counting Task
Description: This outcome is related to the sub-study to investigate the effect of the MBSR on BCI learning. The breath-counting task will be used to measure the participants' mindfulness. Specifically, participants will be asked to count their breaths in cycles of nine (inhale and exhale counting as one) for 18 minutes, pressing one button for the first eight breaths, and a second button for the ninth. Breath counting accuracy is quantified as the number of correctly labeled breath cycles divided by the total number of cycles. The breath-counting accuracy for pre and post-intervention will be used.
Time Frame: 6 months for each participant.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of breath counting accuracy
Arm/Group | Mindfulness Based Stress Reduction - UMN | Waitlist - UMN
Number analyzed (Participants) | 33 | 29
percentage of breath counting accuracy | 93.18 [85.82 to 96.06] | 77.79 [69.40 to 84.59]
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction - UMN vs Waitlist - UMN; Test type: Equivalence — This WRS test will determine if the MBSR group breath counting accuracy was significantly greater than the postintervention levels of controls; p < 0.001, Wilcoxon (Mann-Whitney) — The threshold for statistical analysis was p = 0.05; Mean Difference (Net) = 15.40

3. Primary Outcome: Survey Results and Correlation With BCI Performance
Description: In the first session, participants are asked to complete two surveys to measure one's level of mindfulness before the BCI experiment. In both surveys, a higher score indicates a higher level of mindfulness:
  Survey 1: The Freiburg Mindfulness Inventory (FMI), with 14 statements, such as "I am open to the experience of the present moment". Participants are asked to use a 1-4 scale to indicate how often they have such an experience. The FMI score is calculated by summing up the answers to each question with a proper re-code of one question. FMI score range (minimum to maximum): 14 to 56.
  Survey 2: Day-to-Day Experiences, with 15 questions, such as "I find it difficult to stay focused on what's happening in the present". Participants are asked to use a 1-6 scale to indicate how often they have such an experience. The Mindful Attention Awareness Scale (MAAS) is calculated by averaging answers to each question in this survey. MAAS score range (minimum to maximum): 1 to 6.
Time Frame: During the first experiment session, when each participant did the screening
Population: The population consists of experienced meditators and meditation naive controls. During the analysis, outliers whose BCI performance were outside the ± 2.5 median absolute deviations from the median of the whole sample were excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experienced Meditator - CMU | Meditation Naive - CMU
Number analyzed (Participants) | 14 | 15
score on a scale
  FMI score | 44.5 (4.5) | 36.6 (6.7)
  MAAS score | 4.42 (0.81) | 3.73 (0.67)
Statistical Analysis 1: Comparison: Experienced Meditator - CMU vs Meditation Naive - CMU; Test type: Equivalence — The null hypothesis is that the FMI scores of the two groups have equal medians; p < 0.01, Wilcoxon (Mann-Whitney) — significant if p<0.05; Mean Difference (Final Values) = 7.9
Statistical Analysis 2: Comparison: Experienced Meditator - CMU vs Meditation Naive - CMU; Test type: Equivalence — The null hypothesis is that the MAAS scores of the two groups have equal medians; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.69
Statistical Analysis 3: Comparison: Experienced Meditator - CMU vs Meditation Naive - CMU; Test type: Other — This statistical test is about the correlation between baseline up-down BCI performance and the FMI score. A linear regression model is used to test if the slope is non-zero; p < 0.05, Regression, Linear — significant if p<0.05; correlation coefficient = 0.42
Statistical Analysis 4: Comparison: Experienced Meditator - CMU vs Meditation Naive - CMU; Test type: Other — This statistical test is about the correlation between baseline up-down BCI performance and the MAAS score. A linear regression model is used to test if the slope is non-zero; p < 0.05, Regression, Linear; correlation coefficient = 0.41

ADVERSE EVENTS:
Time Frame: Between when participants were enrolled and completed the last experiment. The period is about 6 months for the sub-study to investigate the effect of MBSR on BCI learning, 1~2 months for the sub-study to investigate the BCI learning of experienced meditators, and 2~3 weeks for the sub-study to examine the effect of short-term meditation on BCI learning.
Arm/Group | Mindfulness Based Stress Reduction - UMN | Waitlist - UMN | Experienced Meditator - CMU | Meditation Naive - CMU | Mindfulness Based Stress Reduction - CMU | Waitlist - CMU | Short Term Meditation - CMU - Meditation | Short Term Meditation - CMU - Control
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72 | 0/32 | 0/34 | 0/8 | 0/8 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/32 | 0/34 | 0/8 | 0/8 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/32 | 0/34 | 0/8 | 0/8 | 0/3 | 0/2

LIMITATIONS AND CAVEATS:
Limitations of the MBSR brain-computer interface sub-study design:

1. The lack of an active control group that requires the same mental commitment of time or intensity as a meditation practice.
2. The exclusive use of the breath counting task as our sole measure of mindfulness.

Limitation of the experienced meditation sub-study design:

Due to the limited sample size, we were unable to determine if the difference in age and sex between groups were significantly influencing the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT03221374/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT03221374/SAP_001.pdf
  • Informed Consent Form (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT03221374/ICF_002.pdf